CLINICAL TRIAL: NCT04530929
Title: Analysis of the Impact of Used Probiotic Strains and Diet on Body Composition, Cardiopulmonary Efficiency and the Incidence of Gastrointestinal Disorders in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Maniac Gym Bialystok (Unknown); University Teaching Hospital, Bialystok (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N/ST/MN/18/003/3316
Record Dates: First submitted 2020-08-10; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Disorder, Functional
Keywords: probiotic; gastrointestinal disorder; long-distance running; body composition; cardiopulmonary efficiency
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: 70 people meeting the inclusion criteria were included in the intervention and observational study. The study was randomized using a double-blind trial. 35 persons selected in the draw were G1 group and the remaining G2 group (n=35). The tests were completely anonymous, the competitors gave their informed written consent to carry them out. Interventional study was conducted using a probiotic or placebo. The intervention factor was the SANPROBI BARRIER multi-strain probiotic (commonly available in pharmacies) or placebo (created on the model of a probiotic capsule, specially for the needs of research, by Sanprobi Sp. z o.o.). Competitors used probiotic/ placebo for three months at a dose of 2x2 capsules daily (2.5 x 109 CFU / g (1 capsule)).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PROBIOTIC (Active Comparator): The intervention factor was the SANPROBI BARRIER multi-strain probiotic (commonly available in pharmacies). Competitors used probiotic for three months at a dose of 2x2 capsules daily (2.5 x 109 CFU / g (1 capsule)).
  Interventions: Dietary Supplement: SANPROBI BARRIER
- Group PLACEBO (Placebo Comparator): Placebo created on the model of a probiotic capsule, specially for the needs of research, by Sanprobi Sp. z o.o.. Competitors used placebo for three months at a dose of 2x2 capsules daily.
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: SANPROBI BARRIER — Competitors used probiotic for three months at a dose of 2x2 capsules daily (2.5 x 109 CFU / g (1 capsule)).
  Arms: Group PROBIOTIC
Dietary Supplement: PLACEBO — Competitors used placebo for three months at a dose of 2x2 capsules daily.
  Arms: Group PLACEBO

SUMMARY:
The aim of the study was to assess the diet and the effect of probiotic therapy on reducing the incidence of gastrointestinal disorders and selected parameters determining the inflammation of the body, body composition, cardiopulmonary efficiency and selected serum biochemical parameters.

70 competitors took part in the study. The research was carried out at the Department of Dietetics and Clinical Nutrition (Medical University of Bialystok), Fitness Club Maniac Gym in Bialystok, as well as at the Hematological Diagnostics Department and the Biochemical Diagnostics Department of the University Teaching Hospital in Bialystok.

The study was randomized using a double-blind trial. 35 persons selected in the draw were G1 group and the remaining G2 group (n=35). The intervention factor was the SANPROBI BARRIER multi-strain probiotic or placebo. Competitors used probiotic/ placebo for three months at a dose of 2x2 capsules daily (2.5 x 10 9 CFU / g (1 capsule)). The consent of the Bioethics Committee of the Medical University, no. RI-002/81/2017, was obtained for the study.

The study consisted of two stages (W1 and W2), and each stage was associated with three visits by the participants. The first of these (W1) included qualification for the study, completing the questionnaire and 3-day nutrition diaries. At the second visit, body composition analysis and cardiopulmonary efficiency test on a medical treadmill were performed. For morphological tests (blood count with smear, lipid profile, fasting glucose, C-reactive protein and ionogram) at the third visit for each competitor was collected blood from the vein in the amount of 10 ml. The final stage (W2) included similar three visits, where the first visit was made after 3 months of taking product A or B. 66 competitors took part in it.

DETAILED DESCRIPTION:
The aim of the study was to assess the diet and the effect of probiotic therapy on reducing the incidence of gastrointestinal disorders and selected parameters determining the inflammation of the body, body composition, cardiopulmonary efficiency and selected serum biochemical parameters.

The approved of the Bioethics Committee of the Medical University, no. RI-002/81/2017, was obtained for the study. 70 people meeting the inclusion criteria were included in the intervention and observational study. The research was carried out at the Department of Dietetics and Clinical Nutrition at the Faculty of Health Sciences of the Medical University of Bialystok, Fitness Club Maniac Gym in Bialystok, as well as at the Hematological Diagnostics Department and the Biochemical Diagnostics Department of the University Clinical Hospital in Bialystok.

The study took place in the spring (March-June 2018) and autumn (September-December 2018), i.e. during of the most intense period in terms of participation in runners' competitions. The study was randomized using a double-blind trial. 35 persons selected in the draw were G1 group and the remaining G2 group (n=35). The tests were completely anonymous, the competitors gave their informed written consent to carry them out.

Interventional study was conducted using a probiotic or placebo. The observation period lasted three months. The intervention factor was the SANPROBI BARRIER multi-strain probiotic (commonly available in pharmacies) or placebo (created on the model of a probiotic capsule, specially for the needs of research, by Sanprobi Sp. z o.o.). Competitors used probiotic/ placebo for three months at a dose of 2x2 capsules daily (2.5 x 10 9 CFU / g (1 capsule)). The probiotic used in the study contained bacterial strains, i.e. Bifidobacterium lactis W52, Lactobacillus brevis W63, Lactobacillus casei W56, Lactococcus lactis W19, Lactococcus lactis W58, Lactobacillus acidophilus W37, Bifidobacterium bifidum W23, Lactobacillus salivarius W24. Players and researchers were not informed about the type of capsule taken (probiotic or placebo). Competitors were asked to use product A or B after blood tests.

Each player had 3 visits during the preliminary stage (W1) and 3 visits of the final stage (W2).

Preliminary stage (W1)

1. The first visit took place in the Department of Dietetics and Clinical Nutrition at the Medical University of Bialystok. It included qualification for the study based on the criteria for inclusion in the study group, discussion of the purpose of the study and signing the written consent for the study by the participants, as well as information about the protection of their personal data and full anonymity. Each participant received an individual code (e.g. A01, A02, B01, B02 etc.), which was used to identify the subject in further stages. Athletes were asked not to use other probiotic strains than those used in the study. All competitors completed a survey regarding demographic data, information on dietary supplementation used, the incidence of gastrointestinal disorders, and 3-day nutrition diary.
2. The second visit took place after a week. Each player was invited to the Maniac Gym Fitness Club in Bialystok. Body composition analysis was performed using an InBody 770 analyzer (InBody, Korea). To determine the level of cardiopulmonary efficiency using the Bruce protocol test on a medical treadmill were performed. Then, competitors were issued a referral for laboratory tests. During this meeting, in accordance with the simple draw product A (group G1) was given to every second person, and product B (group G2) for the remaining persons.
3. For morphological tests (blood count with smear, lipid profile, fasting glucose, C-reactive protein and ionogram) at the third visit for each competitor was collected blood from the vein in the amount of 10 ml.

Final stage (W2) The final stage consisted of three visits (similar to the preliminary stage). The first visit was made after 3 months of taking product A or B by the competitors. 66 people took part in the final stage of the study (G1 = 34 people, G2 = 32 people). One person from group G1 (product A) did not report for the final visit without providing a specific reason. Three people from the G2 control group (product B) did not participate in the final stage of the study (W2) due to injury (2 people) and without providing a specific reason (1 person).

* The first visit took place at the Department of Dietetics and Clinical Nutrition (Medical University of Bialystok) where competitors were completed the questionnaires to determine the changes in the incidence of gastrointestinal disorders.
* The second visit was conducted at the Fitness Club Maniac Gym, where the cardiopulmonary fitness test and body composition analysis were carried out.
* Third visit took place at the Hematological Diagnostics Department of the University Teaching Hospital in Bialystok, where from each participant the blood was collected (from the vein) in an amount of 10 ml for biochemical tests (as during the initial stage at visit 3).

  3-day nutrition diary: Each participant described customary meals consumed for the next three days, including two working days and one day off. The food diary includes hours of meals, the weight of products and dishes, and the amount of fluids consumed during the day. The competitors were asked to use the standard, current diet, without any significant changes. The energy value of the daily nutritional plan, the content of the main nutrients, vitamins, minerals, cholesterol and dietary fiber were taken into account in the evaluation of the three-day nutrition diary. Then, the percentage of compliance with the norm for the energy supply of diet and nutrients was assessed by comparing the results to Polish norms for healthy, adult men and women, and based on scientific research on the discipline of long-distance running.

Body composition analysis All competitors underwent body composition analysis using the InBody model 770 analyzer (South Korea). The body composition analyzer, using the electrical bioimpedance principle, uses low current flow using 6 frequencies and subsequent measurement of the resistance of individual tissues to determine body composition. The following parameters were assessed: body weight (kg), body fat content in kilograms and percent, visceral fat content (cm2), skeletal muscle mass (kg), body water content (kg). Before the test, the participants were informed about the need to stay fasting 8-12 hours and a minimum of 24 hours after physical activity. They were asked to avoid drinking liquids 1 h before the test. None of the competitors had an implanted pacemaker, which is an absolute exclusion criterion in the study of body composition analysis by electrical bioimpedance.

Analysis of cardiopulmonary efficiency In order to determine the cardiopulmonary efficiency of competitors, the Fitmate MED device (Cosmed, Italy) was used, which comprehensively determined cardiopulmonary efficiency and a medical treadmill adapted to this type of HpCosmos analysis (Germany). The Fitmate MED device is equipped with a sensor that enables the measurement of inhaled and exhaled air as well as a mask containing disposable mouthpieces and antibacterial filters. To monitor cardiac contractions, a Garmin sporttester model HRM-Tri 010-10997-09 (United States) was used. In cardiopulmonary fitness tests, a walking treadmill test was used according to Bruce's protocol. The exercise test included effort progression to increase walking speed and incline of the treadmill. The study was divided into 5 stages (3 minutes each). In the first of them, the walk took place at a speed of 2.7 km/h and a 10% incline of the treadmill. In the second stage, the treadmill accelerated to 4 km/h, and the incline increased to 12%. The third stage is a speed of 5.5 km / h and a incline 14%. The fourth stage is the speed increase to 6.8 km / h and the treadmill inclination 16%, and the last stage 5 is the speed of 8 km / h and the inclination of the treadmill 18%. Participants were informed that the cardiorespiratory fitness test should take place for a minimum of 2 weeks after intense physical effort (marathon, ultramarathon). During the test, the maximum test procedure was used to obtain more test parameters, and the test condition was considered to be 90% HRmax by the test subject, or the test could not be continued by interrupting it at the test subject's request. None of the competitors tested completed the test alone, they all reached the 90% HR max limit.

Laboratory tests The tests were performed after venous blood collection (from a vein in the arm) in the amount of 10 ml. Twice (during the initial and final stages) the following measurements were taken: complete blood count with smear, fasting glucose, total cholesterol, HDL, LDL and triglycerides, sodium, iron, potassium, magnesium, serum calcium, determination C-reactive protein (CRP) concentrations. In order to determine pro-inflammatory cytokines, blood was collected on a clot, it was subjected to centrifugation, and after clot separation, the obtained serum was stored at -80 degrees Celsius (until the tests were performed). To determine the concentration of interleukin 6 (IL-6) and tumor necrosis factor (TNF-alpha), the ELISA method (enzyme-linked immunosorbent assay) was used, using R&D System kits (Bio-Techne, United States) according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* women and men aged 20-60,
* running trainings over 5 km/day

Exclusion Criteria:

* use (other than in research) probiotics
* pacemaker

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of probiotic Sanprobi Barrier on the occurrence of gastrointestinal disorders of long-distance runners. | 12 weeks (assessment at baseline and after 3 months of probiotic / placebo use)
  Subjective assessment (survey) of changes in the incidence and severity of gastrointestinal disorders in group of long-distance runners.
  Another survey at the beginning and end of the study.
Influence of probiotic Sanprobi Barrier on the body composition of long-distance runners. | 12 weeks (assessment at baseline and after 3 months of probiotic / placebo use)
  Assessment of runner's body composition changes (body composition analysis used InBody 770 body composition analyzer).
  The following parameters were assessed: body weight (kg), body fat content in kilograms and percent, visceral fat content (cm2), skeletal muscle mass (kg), body water content (kg).
Influence of probiotic Sanprobi Barrier on the cardiopulmonary efficiency of long-distance runners. | 12 weeks (assessment at baseline and after 3 months of probiotic / placebo use)
  Assessment of changes in cardiopulmonary efficiency of long-distance runners (testing the player's efficiency on a medical treadmill with the use of a sport tester and an oxygen mask. Bruce Test Protocol).
Influence of probiotic Sanprobi Barrier on general inflammation of the body. | 12 weeks (assessment at baseline and after 3 months of probiotic / placebo use)
  Assessment of changes in parameters (C-reactive protein, TNF-alpha, IL-6) from blood.
Influence of probiotic Sanprobi Barrier on blood biochemical parameters. | 12 weeks (assessment at baseline and after 3 months of probiotic / placebo use)
  Assessment of changes in parameters (complete blood count with smear, fasting glucose, total cholesterol, HDL, LDL and triglycerides, sodium, iron, potassium, magnesium, serum calcium) from blood.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Smarkusz-Zarzecka, PhD, Principal Investigator — Department of Dietetics and Clinical Nutrition, Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Videbaek S, Bueno AM, Nielsen RO, Rasmussen S. Incidence of Running-Related Injuries Per 1000 h of running in Different Types of Runners: A Systematic Review and Meta-Analysis. Sports Med. 2015 Jul;45(7):1017-26. doi: 10.1007/s40279-015-0333-8. PMID 25951917
- [Background] Vitale K, Getzin A. Nutrition and Supplement Update for the Endurance Athlete: Review and Recommendations. Nutrients. 2019 Jun 7;11(6):1289. doi: 10.3390/nu11061289. PMID 31181616
- [Background] Cox AJ, Pyne DB, Saunders PU, Fricker PA. Oral administration of the probiotic Lactobacillus fermentum VRI-003 and mucosal immunity in endurance athletes. Br J Sports Med. 2010 Mar;44(4):222-6. doi: 10.1136/bjsm.2007.044628. Epub 2008 Feb 13. PMID 18272539
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Huang WC, Lee MC, Lee CC, Ng KS, Hsu YJ, Tsai TY, Young SL, Lin JS, Huang CC. Effect of Lactobacillus plantarum TWK10 on Exercise Physiological Adaptation, Performance, and Body Composition in Healthy Humans. Nutrients. 2019 Nov 19;11(11):2836. doi: 10.3390/nu11112836. PMID 31752370
- [Background] Jager R, Mohr AE, Carpenter KC, Kerksick CM, Purpura M, Moussa A, Townsend JR, Lamprecht M, West NP, Black K, Gleeson M, Pyne DB, Wells SD, Arent SM, Smith-Ryan AE, Kreider RB, Campbell BI, Bannock L, Scheiman J, Wissent CJ, Pane M, Kalman DS, Pugh JN, Ter Haar JA, Antonio J. International Society of Sports Nutrition Position Stand: Probiotics. J Int Soc Sports Nutr. 2019 Dec 21;16(1):62. doi: 10.1186/s12970-019-0329-0. PMID 31864419
- [Background] West NP, Pyne DB, Cripps AW, Hopkins WG, Eskesen DC, Jairath A, Christophersen CT, Conlon MA, Fricker PA. Lactobacillus fermentum (PCC(R)) supplementation and gastrointestinal and respiratory-tract illness symptoms: a randomised control trial in athletes. Nutr J. 2011 Apr 11;10:30. doi: 10.1186/1475-2891-10-30. PMID 21477383
- [Background] Leite GSF, Resende Master Student AS, West NP, Lancha AH Jr. Probiotics and sports: A new magic bullet? Nutrition. 2019 Apr;60:152-160. doi: 10.1016/j.nut.2018.09.023. Epub 2018 Oct 22. PMID 30590242
- [Background] Clark A, Mach N. Exercise-induced stress behavior, gut-microbiota-brain axis and diet: a systematic review for athletes. J Int Soc Sports Nutr. 2016 Nov 24;13:43. doi: 10.1186/s12970-016-0155-6. eCollection 2016. PMID 27924137
- [Background] Holland AM, Hyatt HW, Smuder AJ, Sollanek KJ, Morton AB, Roberts MD, Kavazis AN. Influence of endurance exercise training on antioxidant enzymes, tight junction proteins, and inflammatory markers in the rat ileum. BMC Res Notes. 2015 Sep 30;8:514. doi: 10.1186/s13104-015-1500-6. PMID 26423686
- [Background] Pugh JN, Sparks AS, Doran DA, Fleming SC, Langan-Evans C, Kirk B, Fearn R, Morton JP, Close GL. Four weeks of probiotic supplementation reduces GI symptoms during a marathon race. Eur J Appl Physiol. 2019 Jul;119(7):1491-1501. doi: 10.1007/s00421-019-04136-3. Epub 2019 Apr 13. PMID 30982100
- [Background] Besselink MG, van Santvoort HC, Renooij W, de Smet MB, Boermeester MA, Fischer K, Timmerman HM, Ahmed Ali U, Cirkel GA, Bollen TL, van Ramshorst B, Schaapherder AF, Witteman BJ, Ploeg RJ, van Goor H, van Laarhoven CJ, Tan AC, Brink MA, van der Harst E, Wahab PJ, van Eijck CH, Dejong CH, van Erpecum KJ, Akkermans LM, Gooszen HG; Dutch Acute Pancreatitis Study Group. Intestinal barrier dysfunction in a randomized trial of a specific probiotic composition in acute pancreatitis. Ann Surg. 2009 Nov;250(5):712-9. doi: 10.1097/SLA.0b013e3181bce5bd. PMID 19801929
- [Background] Schmitz L, Ferrari N, Schwiertz A, Rusch K, Woestmann U, Mahabir E, Graf C. Impact of endurance exercise and probiotic supplementation on the intestinal microbiota: a cross-over pilot study. Pilot Feasibility Stud. 2019 Jun 8;5:76. doi: 10.1186/s40814-019-0459-9. eCollection 2019. PMID 31198580
- [Background] Clancy RL, Gleeson M, Cox A, Callister R, Dorrington M, D'Este C, Pang G, Pyne D, Fricker P, Henriksson A. Reversal in fatigued athletes of a defect in interferon gamma secretion after administration of Lactobacillus acidophilus. Br J Sports Med. 2006 Apr;40(4):351-4. doi: 10.1136/bjsm.2005.024364. PMID 16556792
- [Background] West NP, Horn PL, Pyne DB, Gebski VJ, Lahtinen SJ, Fricker PA, Cripps AW. Probiotic supplementation for respiratory and gastrointestinal illness symptoms in healthy physically active individuals. Clin Nutr. 2014 Aug;33(4):581-7. doi: 10.1016/j.clnu.2013.10.002. Epub 2013 Oct 10. PMID 24268677
- [Background] Strasser B, Geiger D, Schauer M, Gostner JM, Gatterer H, Burtscher M, Fuchs D. Probiotic Supplements Beneficially Affect Tryptophan-Kynurenine Metabolism and Reduce the Incidence of Upper Respiratory Tract Infections in Trained Athletes: A Randomized, Double-Blinded, Placebo-Controlled Trial. Nutrients. 2016 Nov 23;8(11):752. doi: 10.3390/nu8110752. PMID 27886064
- [Background] Thomas DT, Erdman KA, Burke LM. Position of the Academy of Nutrition and Dietetics, Dietitians of Canada, and the American College of Sports Medicine: Nutrition and Athletic Performance. J Acad Nutr Diet. 2016 Mar;116(3):501-528. doi: 10.1016/j.jand.2015.12.006. PMID 26920240
- [Background] Jang LG, Choi G, Kim SW, Kim BY, Lee S, Park H. The combination of sport and sport-specific diet is associated with characteristics of gut microbiota: an observational study. J Int Soc Sports Nutr. 2019 May 3;16(1):21. doi: 10.1186/s12970-019-0290-y. PMID 31053143
- [Background] Cartee GD, Hepple RT, Bamman MM, Zierath JR. Exercise Promotes Healthy Aging of Skeletal Muscle. Cell Metab. 2016 Jun 14;23(6):1034-1047. doi: 10.1016/j.cmet.2016.05.007. PMID 27304505
- [Background] Cheng J, Ouwehand AC. Gastroesophageal Reflux Disease and Probiotics: A Systematic Review. Nutrients. 2020 Jan 2;12(1):132. doi: 10.3390/nu12010132. PMID 31906573
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Lamprecht M, Bogner S, Schippinger G, Steinbauer K, Fankhauser F, Hallstroem S, Schuetz B, Greilberger JF. Probiotic supplementation affects markers of intestinal barrier, oxidation, and inflammation in trained men; a randomized, double-blinded, placebo-controlled trial. J Int Soc Sports Nutr. 2012 Sep 20;9(1):45. doi: 10.1186/1550-2783-9-45. PMID 22992437
- [Background] Calero CDQ, Rincon EO, Marqueta PM. Probiotics, prebiotics and synbiotics: useful for athletes and active individuals? A systematic review. Benef Microbes. 2020 Mar 27;11(2):135-149. doi: 10.3920/BM2019.0076. Epub 2020 Feb 19. PMID 32073297
- [Background] Shing CM, Peake JM, Lim CL, Briskey D, Walsh NP, Fortes MB, Ahuja KD, Vitetta L. Effects of probiotics supplementation on gastrointestinal permeability, inflammation and exercise performance in the heat. Eur J Appl Physiol. 2014 Jan;114(1):93-103. doi: 10.1007/s00421-013-2748-y. Epub 2013 Oct 23. PMID 24150782
- [Background] Fedewa MV, Hathaway ED, Ward-Ritacco CL. Effect of exercise training on C reactive protein: a systematic review and meta-analysis of randomised and non-randomised controlled trials. Br J Sports Med. 2017 Apr;51(8):670-676. doi: 10.1136/bjsports-2016-095999. Epub 2016 Jul 21. PMID 27445361
- [Background] Huang WC, Wei CC, Huang CC, Chen WL, Huang HY. The Beneficial Effects of Lactobacillus plantarum PS128 on High-Intensity, Exercise-Induced Oxidative Stress, Inflammation, and Performance in Triathletes. Nutrients. 2019 Feb 7;11(2):353. doi: 10.3390/nu11020353. PMID 30736479
- [Background] Wosinska L, Cotter PD, O'Sullivan O, Guinane C. The Potential Impact of Probiotics on the Gut Microbiome of Athletes. Nutrients. 2019 Sep 21;11(10):2270. doi: 10.3390/nu11102270. PMID 31546638
- [Background] Kim J, Yun JM, Kim MK, Kwon O, Cho B. Lactobacillus gasseri BNR17 Supplementation Reduces the Visceral Fat Accumulation and Waist Circumference in Obese Adults: A Randomized, Double-Blind, Placebo-Controlled Trial. J Med Food. 2018 May;21(5):454-461. doi: 10.1089/jmf.2017.3937. Epub 2018 Apr 24. PMID 29688793
- [Derived] Smarkusz-Zarzecka J, Ostrowska L, Leszczynska J, Cwalina U. Effect of a Multi-Strain Probiotic Supplement on Gastrointestinal Symptoms and Serum Biochemical Parameters of Long-Distance Runners: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Jul 30;19(15):9363. doi: 10.3390/ijerph19159363. PMID 35954716